CLINICAL TRIAL: NCT03622554
Title: Strengthening Equilibrium and Educational Support in Preventing Falls in the Thermal Center
Acronym: RESPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Association Francaise pour la Recherche Thermale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UF7664
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Prevention of Falls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Curist taking a spa treatment of 3 weeks in the usual conditions for each Center
- Intervention (Experimental): Addition to the usual cure: -12 adapted physical activity (APA) sessions of 60 minutes to improve the balance , muscular strength, endurance and suppleness without creating additional fatigue for the curists
  - personalized therapeutic patient education (ETP) with an individual assessment at the beginning of the treatment (1h), 3 group sessions (1h30) and an end-of-cure interview (1h) and an educational follow-up by phone at 3, 6 and 12 months
  Interventions: Other: Adapted Physical Activity (APA); Other: Therapeutic Patient Education (ETP)

INTERVENTIONS:
Other: Adapted Physical Activity (APA) — 12 APA sessions of 60 minutes
  Arms: Intervention
Other: Therapeutic Patient Education (ETP) — Personalized ETP with 3 group sessions (1h30) and one at the end of the course (1h) and educational follow-up by phone at 3, 6 and 12 months
  Arms: Intervention

SUMMARY:
Preventing falls among people 65 years of age or older is a priority to promote healthy aging and reduce the number of hospitalizations, institutionalizations and years lived with disability. A preliminary study carried out at the Balaruc-les-Bains Thermal Center showed that one-third of people aged 65 are at significant risk of falling. Thermal establishments could therefore play a role in initiating measures to prevent falls among people aged 65 and over screened at risk.The main objective is to evaluate the impact on the incidence of falls at 12 months (M12) to add to the usual care (control group) a program combining, during the treatment, adapted physical activities (APA) and a Therapeutic patient education (FTE) followed by an educational follow-up for 12 months (intervention group) for people aged 65 and over who were at risk of falling on arrival at the Thermal

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 65 and over,
* Presence of at least one chronic pathology justifying treatment and cure
* Subject having a history of fall in the last year (at least one fall)
* Subject having at least one risk factor of falling among the following 3: balance disorder, decreased muscle strength or gait disorder

Exclusion Criteria:

* Subject considered by the investigators as not being able to participate in the program (inability to answer questionnaires, to perform tests, for example).
* Patient under the protection of justice, under guardianship or curatorship

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 269 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Incidence of falls at 12 months | 12 months
  To evaluate the impact on the incidence of falls at 12 months (M12) to add to the usual care (control group) a program combining, during the treatment, adapted physical activities (APA) and therapeutic patient education ( ETP), followed by an educational follow-up for 12 months (intervention group) for people aged 65 and over who were at risk of falling on arrival at the Thermal Center

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No